CLINICAL TRIAL: NCT03740867
Title: Does Cognitive Status Affect Pulmonary Rehabilitation Gains?
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, esra pehlivan, Principal investigator, Istanbul Medipol University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Cognition_PR
Record Dates: First submitted 2018-11-02; First posted 2018-11-14 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Cognitive Impairment; Pulmonary Rehabilitation
Keywords: Cognitive Impairment; pulmonary rehabilitation; exercise; MOCA; aerobic training
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Intervention Model Description: After completion of the program, patients will be divided into two groups according to their cognitive status (Group 1: those with poor cognition; Group 2: those with good cognition). The PR gains of the groups will be compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1 (Experimental): Those with poor cognition (MOCA score<23)
  The patients will receive the Pulmonary Rehabilitation program for 3-months (2 days at hospital, 3 days at home). Exercise program includes aerobic (walking band, bicycle, arm ergometer) and strengthening (with free weights) components.
  Interventions: Other: Pulmonary rehabilitation
- Group2 (Experimental): Those with good cognition (MOCA score≥23)
  The patients will receive the Pulmonary Rehabilitation program for 3-months (2 days at hospital, 3 days at home). Exercise program includes aerobic (walking band, bicycle, arm ergometer) and strengthening (with free weights) components.
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Pulmonary rehabilitation — Exercise program includes aerobic (walking band, bicycle, arm ergometer) and strengthening (with free weights) components.

SUMMARY:
Pulmonary rehabilitation program with aerobic and strengthening trainings for 3 months will be applied to the candidates for lung transplantation. The program will be designed to be 2 days supervised weekly and 3 day home program. After completion of the program, patients will be divided into two groups according to their cognitive status (Group 1: those with poor cognition; Group 2: those with good cognition). The PR gains of the groups will be compared.

DETAILED DESCRIPTION:
The fact that cognition is not always included in the assessment routine makes it difficult to clarify which patient group or severity of illness is more affected by this issue. The effect of exercise on cognitive functions is a remarkable issue in recent years. It can also be predicted that cognitive function may be effective on program adaptation in patients who are given home program without supervision. The aim of the investigator's study was to investigate the effect of cognitive status to pulmonary rehabilitation gains in lung transplant candidates.

Lung transplantation candidates who refered from Lung Transplantation surgery team will receive the Pulmonary Rehabilitation program for 3-months (2 days at hospital, 3 days at home). Exercise program includes aerobic (walking band, bicycle, arm ergometer) and strengthening (with free weights) components. Patient will evaluate at the beginning and end of the program. Demographic information, diagnosis distributions, educational status of patients will be recorded. Exercise capacities are determined by 6 min walk test. The medical research council dyspnea scale is used in determining the dispense levels. Montreal Cognitive Function Assessment (MOCA) is used to determine cognitive functions. Cognitive functions and exercise capacities of the patients before and after the program will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* To be listed for lung transplantation,
* Pulmonary rehabilitation exercise program planned to be taken,
* Volunteers who have agreed to participate in the work,
* Patients who can complete the 3-month Pulmonary Rehabilitation program.

Exclusion Criteria:

* Failure to complete the planned exercise program for any reason,
* Not to be literate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-11-13 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline the 6 minutes walk distance at 3 months. | 3 months
  The test was conducted in a 30-m corridor in line with American Thoracic Society (ATS) guidelines. Patients were told that they should walk as fast as they can walk in 6 minutes time.
Change from Baseline the Montreal Cognitive Assessment (MoCA) test score at 3 months. | 3 months
  It was designed to detect mild cognitive impairment.Thirty items assessing multiple cognitive domains are contained in the MoCA: short-term memory (5 points); visuospatial abilities via clock drawing (3 points), and a cube copy task (1 point); executive functioning via an adaptation of Trail Making Test Part B (1 point), phonemic fluency (1 point), and verbal abstraction (2 points); attention, concentration, and working memory via target detection (1 point), serial subtraction (3 points), digits forward (1 point), and digits backward (1 point); language via confrontation naming with low-familiarity animals (3 points), and repetition of complex sentences (2 points); and orientation to time and place (6 points). The MoCA is scored by obtaining an item total and the authors recommend a clinical cutoff score of 23.

SECONDARY OUTCOMES:
Change from Baseline the modified Medical Council Dyspnea score at 3 months. | 3 months
  The scale will rate the sensation of dyspnea as the person perceives it.The severity of dyspnea is rated on a scale of 0 to 4."0 point" means no dyspnea perception and "4point" means severe dyspnea perception.
Change from Baseline the Forced Expiratory Volume in 1 second (FEV1) at 3 months. | 3 months
  It was conducted using the Sensor Medics model 2400 (Yorba Linda, CA,USA), according to the ATS guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Pehlivan, PhD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Yedikule Chest Disease Hospital, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided